CLINICAL TRIAL: NCT07310511
Title: Emotional Regulation & Addiction : Impact of In-person/Online Dialectic Behavior Therapy (DBT) vs Usual Treatment
Acronym: RégulAddict
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RC25-0041
Record Dates: First submitted 2025-12-04; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Addiction Disorders; Emotional Dysregulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with emotional dysregulation treated by face-to-face DBT (Experimental)
  Interventions: Behavioral: Face-to-face DBT
- Patients with emotional dysregulation treated by online DBT (Experimental)
  Interventions: Behavioral: Online DBT
- Patients with emotional dysregulation treated by usual treatment (Active Comparator)
  Interventions: Behavioral: Usual treatment

INTERVENTIONS:
Behavioral: Face-to-face DBT — One therapy session per week for two 3-month periods, to learn and practice emotional regulation skills.
  Arms: Patients with emotional dysregulation treated by face-to-face DBT
Behavioral: Online DBT — Two 3-months periods, consisting of watching a video on an emotional regulation skill and completing a worksheet related to that skill. In addition, participants will be encouraged to regularly use mobile apps on emotional regulation.
  Arms: Patients with emotional dysregulation treated by online DBT
Behavioral: Usual treatment — Consultations in the addiction treatment department at a frequency deemed clinically necessary by the professional providing follow-up care. Occupational group therapy (discussion groups, writing, etc.) is usually offered to patients, who may participate as they wish.
  Arms: Patients with emotional dysregulation treated by usual treatment

SUMMARY:
In psychiatry, psychotherapy is, along with pharmacotherapy, a major therapeutic intervention. It helps patients better understand their difficulties and informs them of possible solutions. It is systematically recommended in cases of psychiatric disorders, whether or not in combination with pharmacotherapy.

With regard to addictive disorders in particular, few medications are available and psychotherapy is essential. Psychotherapy must be adapted to the severity of the patient's condition and the issues encountered. In cases of impaired emotional regulation, i.e., the ability to respond effectively to one's emotions, addictions become more difficult to stabilize without appropriate treatment. For patients with emotional regulation disorders, Dialectical Behavior Therapy (DBT) is the standard treatment. It consists of teaching acceptance and change skills in a dialectical manner to better regulate emotions.

Like other evidence-based psychotherapies, DBT is nevertheless not widely available. It requires therapists to have a high level of training and sufficient patient recruitment to form groups. Two solutions are being considered to improve the accessibility of DBT. To facilitate patient recruitment, transdiagnostic groups are useful because they bring together patients with different diagnoses. To help professionals deliver the therapy, digital tools such as pre-recorded videos or mobile applications have proven effective, particularly when guided by a therapist, but they also show some effectiveness without a therapist. Studies are still recent and few in number, and need to be replicated, particularly using a variety of digital tools.

The investigators want to evaluate the effectiveness of DBT on emotional regulation and impulsivity in addiction patients, in a transdiagnostic face-to-face format and in an online format using videos, compared to a control group (usual treatment). This research would provide a better understanding of the effectiveness of DBT in addiction treatment, as well as the effectiveness of solutions that improve its accessibility, such as the transdiagnostic format and the use of associated digital tools.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years
* Patients affiliated with a social security health insurance plan
* Patients who are fluent in French, able to understand the objectives and risks associated with the research, and able to give dated and signed informed consent
* Patients with addictive disorders (substance and/or behavioral) presenting emotional dysregulation (DERS score >90) in the 3 months prior to the inclusion visit
* Patients whose treatment(s) for mood disorder regulation has been stable for 3 months
* No ongoing structured psychotherapy

Exclusion Criteria:

* Patients diagnosed with acute psychosis
* Patients with major neurocognitive disorders
* Patients with encephalopathy
* Patients in a period of exclusion (determined by a previous or ongoing study)
* Patients in an emergency/life-threatening situation
* Patients under legal protection
* Pregnancy (self-reported)/breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Score on the Difficulties in Emotion Regulation Scale (DERS) measured at the first post-therapy follow-up visit (visit V2) in the face-to-face DBT group ant the control group | Between Day 90 and Day 150

CONTACTS AND LOCATIONS:
Overall Officials: Amaury Durpoix, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No